CLINICAL TRIAL: NCT00730938
Title: The Effect of Intracameral Cefuroxime on Post-op Fibrin in Pediatric Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Presbyterian Church East Africa Kikuyu Hospital (Other)
Responsible Party: Dan Gradin, MD, Presbyterian Church East Africa Kikuyu Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kikuyu01
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Cataract; Endophthalmitis
Keywords: fibrin; endophthalmitis; cataract extraction; Lens; implantation,; intraocular
MeSH Terms: conditions — Cataract; Endophthalmitis | interventions — Cefuroxime; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: cefuroxime
- 2 (Placebo Comparator): Saline placebo
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Drug: cefuroxime — intracameral cefuroxime 0.1 ml
  Other Names: Zinacef
  Arms: 1
Drug: Saline placebo — 0.1 ml of Ringers lactate
  Other Names: Saline
  Arms: 2

SUMMARY:
The study investigates whether placing an antibiotic inside the eye at the end of cataract surgery in children will reduce the amount of fibrin formation (fibrin formation can block the pupil and reduce vision). We hypothesize that the fibrin is caused by a low-level infection and could be prevented by the antibiotic.

DETAILED DESCRIPTION:
The study investigates whether using an antibiotic (cefuroxime) in the anterior chamber of the eye at the end of surgery for cataract in children will reduce the amount of fibrin formation.

ELIGIBILITY:
Inclusion Criteria:

* bilateral congenital or developmental pediatric cataract

Exclusion Criteria:

* traumatic cataract

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Fibrin formation in anterior chamber | 4th postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Dan Gradin, MD, Principal Investigator — PCEA Kikuyu Hospital
Locations (1):
- Presbyterian Church East Africa Kikuyu Hospital, Kikuyu, Kenya

REFERENCES:
- [Derived] Gradin D, Mundia D. Effect of intracameral cefuroxime on fibrinous uveitis after pediatric cataract surgery. J Pediatr Ophthalmol Strabismus. 2011 Jan-Feb;48(1):45-9. doi: 10.3928/01913913-20100420-03. Epub 2010 Apr 22. PMID 20438039